CLINICAL TRIAL: NCT00322439
Title: Observational Post-Marketing Safety Surveillance Registry of Enbrel (Etanercept) for Treatment of Psoriasis
Brief Title: Observational Safety Study of Etanercept (Enbrel) for Treatment of Psoriasis
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20040210
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Psoriasis
Keywords: plaque Psoriasis patients; TNF-inhibitor naïve
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Etanercept: Participants received etanercept (Enbrel) treatment at the dose and regimen determined by the investigator and were evaluated for up to 5 years at 6-month intervals. During this period, participants may have discontinued etanercept therapy, may have switched to another anti-psoriatic therapy, may have used etanercept in combination with other anti-psoriatic therapies, or may have discontinued any or all antipsoriatic treatments.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Observational study - no drug administered

SUMMARY:
This is an observational safety study tracking psoriasis patients on etanercept (Enbrel) for 5 years.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational surveillance registry to evaluate data on the long-term safety of etanercept (Enbrel) use in the treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque psoriasis

Exclusion Criteria:

* Prior exposure to any tumor necrosis factor (TNF)-inhibitor
* Patients for whom Enbrel is contraindicated
* Patients currently enrolled in or has not yet completed at least 30 days since ending other investigational drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with plaque psoriasis, who are currently receiving Enbrel or who are intending to start or restart Enbrel therapy at multi-centers.
Sampling Method: Probability Sample
Enrollment: 2511 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2012-12-11 (Actual); Study Completion 2013-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Kimball AB, Pariser D, Yamauchi PS, Menter A, Teller CF, Shi Y, Creamer K, McCroskery P, Kricorian G, Gelfand JM. OBSERVE-5, an Observational Post-Marketing SafetySurveillance Registry of Etanercept for the treatment of Psoriasis: A Model for Studying New Psoriasis Therapies. Psoriasis Forum. 2010;16(3):3-7.
- [Background] Kimball AB, Pariser D, Yamauchi PS, Menter A, Teller CF, Shi Y, Yong M, Creamer K, Hooper M, Aras G, Kricorian G, Gelfand JM. OBSERVE-5 interim analysis: an observational postmarketing safety registry of etanercept for the treatment of psoriasis. J Am Acad Dermatol. 2013 May;68(5):756-64. doi: 10.1016/j.jaad.2012.10.055. Epub 2013 Jan 26. PMID 23357569
- [Background] Kimball AB, Rothman KJ, Kricorian G, Pariser D, Yamauchi PS, Menter A, Teller CF, Aras G, Accortt NA, Hooper M, Rice KC, Gelfand JM. OBSERVE-5: observational postmarketing safety surveillance registry of etanercept for the treatment of psoriasis final 5-year results. J Am Acad Dermatol. 2015 Jan;72(1):115-22. doi: 10.1016/j.jaad.2014.08.050. Epub 2014 Sep 26. PMID 25264239
- [Background] Kimball AB, Schenfeld J, Accortt NA, Anthony MS, Rothman KJ, Pariser D. Incidence rates of malignancies and hospitalized infectious events in patients with psoriasis with or without treatment and a general population in the U.S.A.: 2005-09. Br J Dermatol. 2014 Feb;170(2):366-73. doi: 10.1111/bjd.12744. PMID 24251402
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etanercept
Started | 2511
Received at Least 1 Dose of Etanercept | 2510
Completed | 1455
Not Completed | 1056

BASELINE CHARACTERISTICS:
Population: Full Analysis Set, which consisted of all participants who received at least one dose of etanercept during the study.
Arm/Group | Etanercept
Number analyzed (Participants) | 2510
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.32 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1193
  Male | 1317
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 2052
  Black or African American | 108
  Hispanic or Latino | 164
  Asian | 116
  Japanese | 4
  American Indian or Alaska Native | 8
  Native Hawaiian or Other Pacific Islander | 23
  Other | 35

OUTCOME MEASURES:

1. Primary Outcome: Five-year Cumulative Incidence of Serious Adverse Events and Serious Infectious Events
Description: A serious adverse event (SAE), including a serious infectious event (SIE), is defined as one that suggests a significant hazard or side effect, regardless of the investigator or sponsor's opinion on the relationship to a drug product. This includes, but may not be limited to, any event that (at any dose) is fatal, life threatening, requires inpatient hospitalization that includes a minimum of an overnight stay or prolongation of existing hospitalization, is a persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. Cumulative incidences were calculated using Kaplan-Meier methodology for all participants who received at least 1 registry dose of etanercept. For SAEs and SIEs, time to event was re-defined from calendar time to cumulative time up to the event, excluding time intervals and events when the participant was not on etanercept treatment (ie, based on etenercept exposure time).
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 2510
proportion of participants
  Serious Adverse Events | 0.2029 [0.1799 to 0.2260]
  Serious Infectious Events | 0.0581 [0.0447 to 0.0716]

2. Secondary Outcome: Five-year Cumulative Incidence for Events of Medical Interest (EMIs)
Description: Protocol defined EMIs included: • All malignancies, including basal cell carcinoma (BCC) and squamous cell carcinoma (SCC); • Tuberculosis; • Opportunistic infections treated with intravenous therapy; • Histoplasmosis infections treated with oral antibiotics; • Coccidioidomycosis infections treated with oral antibiotics; • Central nervous system (CNS) demyelinating disorders; • Lupus disease; • Coronary artery disease; • Worsening of psoriasis as defined by change in psoriasis morphology and withdrawal of therapy; • Any event or laboratory abnormality that represents an event of medical significance. Cumulative incidences were calculated using Kaplan-Meier methods where time to event was defined as the time from the first dose of etanercept to the start date of the first occurrence of the event, regardless of exposure (ie, based on observation time). Estimates were adjusted using left truncation methodology to help address any bias due to participants with prior etanercept exposure.
Time Frame: 5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 2510
proportion of participants
  Malignancy, including BCC, SCC and lymphoma | 0.0659 [0.0538 to 0.0780]
  Coronary artery disease | 0.0283 [0.0202 to 0.0364]
  Worsening of psoriasis | 0.0074 [0.0032 to 0.0115]
  CNS demyelinating disorder | 0.0018 [-0.0002 to 0.0039]
  Tuberculosis | 0.0013 [-0.0005 to 0.0030]
  Lupus disease | 0.0006 [-0.0006 to 0.0018]
  Opportunistic infection | 0.0006 [-0.0006 to 0.0018]
  Coccidioidomycosis | NA [NA to NA] — There were no events in this category
  Histoplasmosis | NA [NA to NA] — There were no events in this category

3. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) of Psoriasis Score of 0 (Clear) or 1 (Almost Clear)
Description: The sPGA scale is designed to evaluate the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA is assessed on a scale of 0 to 5 (0 = clear, 5 = severe).
Time Frame: Baseline and at 3 and 5 years
Population: Participants who received at least one registry dose of etanercept, excluding participants who were enrolled at sites that were closed for cause, and with available data at each time point (indicated by n).
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
percentage of participants
  Baseline (n=2472) | 12.0
  3 years (n= 1456) | 47.4
  5 years (n=1269) | 51.5

4. Secondary Outcome: Percentage of Participants With a Patient's Global Assessment of Psoriasis Score of 0 or 1
Description: The patient's global assessment of psoriasis is a self-administered numeric scale is designed to evaluate participants' perception of their psoriasis on a scale from 0 (good) to 5 (severe).
Time Frame: Baseline and at 3 and 5 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
percentage of participants
  Baseline (n=2435) | 11.4
  3 years (n= 1446) | 53.2
  5 years (n=1322) | 55.7

5. Secondary Outcome: Percentage of Participants With a Dermatology Life Quality Index (DLQI) Response
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. A DLQI response is defined as a 5 point improvement from Baseline or a score of 0.
Time Frame: Baseline, Year 3 and Year 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
percentage of participants
  Year 3 (n=1453) | 60.2
  Year 5 (n=1319) | 64.5

6. Secondary Outcome: Euroqol-5D (EQ-5D) Total Score
Description: EQ-5D is a self-reported questionnaire that consists of five single-item health domains, mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers are recorded as choices of 1, 2, or 3 for each question, with 1 signifying no problem, 2 signifying some problem, and 3 signifying major problem. Using the US scoring algorithm, the possible total EQ-5D score ranges from -0.11 (ie, answered '3' for all questions) to 1.0 (ie, answered '1' for all questions), where 1.0 represents perfect health.
Time Frame: Baseline, Year 3 and Year 5
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
units on a scale
  Baseline (n=2440) | 0.78 (0.0)
  Year 3 (n=1454) | 0.86 (0.0)
  Year 5 (n=1322) | 0.86 (0.0)

7. Secondary Outcome: Euroqol-5D (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D visual analog scale (VAS) is a 100 mm scale with 100 representing 'best imaginable health state' and 0 representing 'worst imaginable health state'. Participants were asked to indicate on this scale how good or bad their health was today.
Time Frame: Baseline, Year 3 and Year 5
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
units on a scale
  Baseline (n=2446) | 74.05 (0.40)
  Year 3 (n=1462) | 81.81 (0.42)
  Year 5 (n=1328) | 82.51 (0.44)

8. Secondary Outcome: Healthcare Resource Use
Description: This self-administered questionnaire is designed to measure the amount of healthcare resource utilization by the participant in the past 4 weeks. The average answers to the following questions are reported:
  1. How many times have you been to any physician's office or urgent care clinic, not including your dermatologist?
  2. How many times have you seen a nurse practitioner, physician assistant, psychologist, naturopath, acupuncturist, or chiropractor?
  3. How many times have you received care from a health professional (HP) in your home?
  4. How many times have you paid someone to help you do chores around the house (cleaning, maintenance, lawn care)?
  5. How many times have you had a friend or family member take time off work to provide care or transportation?
Time Frame: Baseline, Year 3 and Year 5
Population: as for outcome 3
Measure: Mean (Standard Error); unit: times
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
times
  Baseline: Physician/urgent care visits (n=2423) | 0.72 (0.0)
  Baseline: Nurse practitioner, etc visits (n=2418) | 0.35 (0.0)
  Baseline: Home care from a HP (n=2411) | 0.03 (0.0)
  Baseline: Paid help with chores (n=2414) | 0.46 (0.0)
  Baseline: Friend or family provided care (n=2415) | 0.26 (0.0)
  Year 3: Physician/urgent care visits (n=1458) | 0.63 (0.0)
  Year 3: Nurse practitioner, etc visits (n=1451) | 0.29 (0.0)
  Year 3: Home care visits from a HP (n=1451) | 0.03 (0.0)
  Year 3: Paid help with chores (n=1451) | 0.42 (0.0)
  Year 3: Friend or family provided care (n=1453) | 0.12 (0.0)
  Year 5: Physician/urgent care visits (n=1317) | 0.64 (0.0)
  Year 5: Nurse practitioner, etc visits (n=1318) | 0.27 (0.0)
  Year 5: Home care visits from a HP (n=1317) | 0.06 (0.0)
  Year 5: Paid help with chores (n=1318) | 0.44 (0.1)
  Year 5: Friend or family provided care (n=1318) | 0.17 (0.0)

9. Secondary Outcome: Work Productivity and Activity Impairment (WPAI)
Description: The WPAI questionnaire has six questions to assess whether the participant was currently employed (Q1); how many hours from work were missed due to problems associated with psoriasis (Q2) or any other reason (Q3); hours actually worked (Q4); degree that psoriasis affected productivity while working (Q5); and degree that psoriasis affected regular activities (Q6) over the past 7 days. Four separate overall scores were calculated, including absenteeism (work time missed due to health), presenteeism (impairment at work due to health), work productivity loss (overall work impairment due to health), and activity impairment due to health. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity (ie, worse outcomes).
Time Frame: Baseline, Year 3 and Year 5
Population: Participants who received at least one registry dose of etanercept, excluding participants who were enrolled at sites that were closed for cause, and with available data at each time point (indicated by n), and who were employed (for the first 3 scores).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
units on a scale
  Absenteeism - Baseline (n=1709) | 2.81 (0.28)
  Absenteeism - Year 3 (n=949) | 1.34 (0.23)
  Absenteeism - Year 5 (n=808) | 1.47 (0.32)
  Presenteeism - Baseline (n=1832) | 18.50 (0.57)
  Presenteeism - Year 3 (n=1009) | 9.00 (0.59)
  Presenteeism - Year 5 (n=866) | 7.90 (0.58)
  Work Productivity Loss - Baseline (n=1702) | 18.82 (0.60)
  Work Productivity Loss - Year 3 (n=944) | 9.58 (0.63)
  Work Productivity Loss - Year 5 (n=805) | 8.55 (0.65)
  Activity Impairment - Baseline (n=2440) | 25.37 (0.57)
  Activity Impairment - Year 3 (n=1460) | 12.01 (0.55)
  Activity Impairment - Year 5 (n=1322) | 11.29 (0.57)

10. Secondary Outcome: Percentage of Body Surface Area Affected by Psoriasis
Description: Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis.
Time Frame: Baseline, Year 3 and Year 5
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Etanercept
Number analyzed (Participants) | 2493
percentage of body surface area
  Baseline (n=2478) | 21.06 (0.39)
  Year 3 (n=1455) | 6.59 (0.28)
  Year 5 (n=1269) | 6.06 (0.30)

ADVERSE EVENTS:
Time Frame: 5 years
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 418/2510
Other Adverse Events (participants affected / at risk) | 0/2510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=2510)
Anaemia (Blood and lymphatic system disorders) | 3
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 3
Acute Myocardial Infarction (Cardiac disorders) | 3
Angina Pectoris (Cardiac disorders) | 8
Angina Unstable (Cardiac disorders) | 1
Aortic Valve Disease (Cardiac disorders) | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 8
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 2
Cardiac Failure Congestive (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 14
Coronary Artery Insufficiency (Cardiac disorders) | 1
Coronary Artery Occlusion (Cardiac disorders) | 2
Coronary Artery Stenosis (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Heart Valve Incompetence (Cardiac disorders) | 1
Mitral Valve Incompetence (Cardiac disorders) | 1
Mitral Valve Prolapse (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 17
Palpitations (Cardiac disorders) | 1
Adrenoleukodystrophy (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Autoimmune Thyroiditis (Endocrine disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Ophthalmoplegia (Eye disorders) | 1
Visual Acuity Reduced (Eye disorders) | 1
Abdominal Adhesions (Gastrointestinal disorders) | 1
Abdominal Hernia (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 2
Alcoholic Pancreatitis (Gastrointestinal disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Crohn's Disease (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Diverticulum Gastric (Gastrointestinal disorders) | 1
Faeces Discoloured (Gastrointestinal disorders) | 1
Gastric Volvulus (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4
Hiatus Hernia (Gastrointestinal disorders) | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 6
Pancreatitis Acute (Gastrointestinal disorders) | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 4
Umbilical Hernia (Gastrointestinal disorders) | 2
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest Discomfort (General disorders) | 2
Chills (General disorders) | 1
Cyst (General disorders) | 1
Death (General disorders) | 17
Device Malfunction (General disorders) | 1
Generalised Oedema (General disorders) | 1
Injection Site Urticaria (General disorders) | 1
Medical Device Complication (General disorders) | 1
Multi-Organ Failure (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 5
Oedema (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 5
Biliary Dyskinesia (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 8
Cholecystitis Acute (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 2
Chronic Hepatic Failure (Hepatobiliary disorders) | 2
Cirrhosis Alcoholic (Hepatobiliary disorders) | 2
Hepatic Cirrhosis (Hepatobiliary disorders) | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 2
Hepatitis Alcoholic (Hepatobiliary disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Abdominal Abscess (Infections and infestations) | 1
Abscess Intestinal (Infections and infestations) | 1
Abscess Limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 4
Arteriovenous Graft Site Infection (Infections and infestations) | 1
Beta Haemolytic Streptococcal Infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 22
Chest Wall Abscess (Infections and infestations) | 1
Cholecystitis Infective (Infections and infestations) | 1
Clostridial Infection (Infections and infestations) | 2
Clostridium Difficile Colitis (Infections and infestations) | 1
Clostridium Difficile Sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 11
Dural Abscess (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia Infection (Infections and infestations) | 1
Escherichia Sepsis (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Hepatitis C (Infections and infestations) | 2
Herpes Zoster (Infections and infestations) | 4
Infectious Mononucleosis (Infections and infestations) | 1
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Injection Site Cellulitis (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 2
Klebsiella Bacteraemia (Infections and infestations) | 1
Latent Tuberculosis (Infections and infestations) | 2
Liver Abscess (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Meningitis Aseptic (Infections and infestations) | 2
Meningitis Listeria (Infections and infestations) | 1
Meningitis Streptococcal (Infections and infestations) | 1
Necrotising Fasciitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Pelvic Inflammatory Disease (Infections and infestations) | 1
Perirectal Abscess (Infections and infestations) | 1
Peritonitis Bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 30
Pneumonia Bacterial (Infections and infestations) | 2
Pneumonia Staphylococcal (Infections and infestations) | 1
Post Procedural Infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 5
Septic Shock (Infections and infestations) | 1
Staphylococcal Abscess (Infections and infestations) | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 7
Subcutaneous Abscess (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 1
Toxic Shock Syndrome (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 2
Viral Infection (Infections and infestations) | 1
Wound Infection Staphylococcal (Infections and infestations) | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1
Crushing Injury Of Trunk (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Femur Fracture (Injury, poisoning and procedural complications) | 1
Foot Fracture (Injury, poisoning and procedural complications) | 3
Fractured Sacrum (Injury, poisoning and procedural complications) | 1
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 3
Injury (Injury, poisoning and procedural complications) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Joint Injury (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 2
Muscle Strain (Injury, poisoning and procedural complications) | 1
Nail Injury (Injury, poisoning and procedural complications) | 1
Patella Fracture (Injury, poisoning and procedural complications) | 2
Pelvic Fracture (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 5
Road Traffic Accident (Injury, poisoning and procedural complications) | 5
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 2
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1
Traumatic Renal Injury (Injury, poisoning and procedural complications) | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Ureteric Injury (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Anticonvulsant Drug Level Increased (Investigations) | 1
Antinuclear Antibody Positive (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Lipase Increased (Investigations) | 1
Tuberculin Test Positive (Investigations) | 1
White Blood Cell Count Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Diabetes Mellitus (Metabolism and nutrition disorders) | 3
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2
Failure To Thrive (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Obesity (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 8
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 5
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B Precursor Type Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Uterine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Large Cell Carcinoma Of The Respiratory Tract Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mycosis Fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Oesophageal Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Precursor B-Lymphoblastic Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Rectal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arachnoid Cyst (Nervous system disorders) | 1
Arachnoiditis (Nervous system disorders) | 1
Balance Disorder (Nervous system disorders) | 1
Benign Intracranial Hypertension (Nervous system disorders) | 1
Carotid Artery Occlusion (Nervous system disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 4
Dementia (Nervous system disorders) | 1
Diabetic Neuropathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hepatic Encephalopathy (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Intracranial Aneurysm (Nervous system disorders) | 1
Intracranial Pressure Increased (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 1
Loss Of Consciousness (Nervous system disorders) | 1
Multiple Sclerosis (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 2
Parkinson's Disease (Nervous system disorders) | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Radicular Syndrome (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Thoracic Outlet Syndrome (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 4
Complication Of Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1
Adjustment Disorder With Mixed Disturbance Of Emotion And Conduct (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bipolar Disorder (Psychiatric disorders) | 2
Completed Suicide (Psychiatric disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Major Depression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Psychotic Disorder (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Suicide Attempt (Psychiatric disorders) | 1
Calculus Ureteric (Renal and urinary disorders) | 1
Glomerulonephritis Membranous (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 7
Renal Aneurysm (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 4
Renal Failure Acute (Renal and urinary disorders) | 6
Renal Failure Chronic (Renal and urinary disorders) | 4
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Ovarian Mass (Reproductive system and breast disorders) | 1
Polycystic Ovaries (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Uterine Polyp (Reproductive system and breast disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2
Caesarean Section (Surgical and medical procedures) | 2
Aortic Aneurysm (Vascular disorders) | 1
Aortic Dissection (Vascular disorders) | 2
Arteriosclerosis (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 5
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2
Intermittent Claudication (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
Peripheral Vascular Disorder (Vascular disorders) | 1
Superior Vena Cava Syndrome (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.